CLINICAL TRIAL: NCT00154024
Title: Characterization of Local Vascular Effects of Angiotensin II and Histamine After Treatment With Irbesartan and Atorvastatin.
Brief Title: Comparison of Vascular Effects After Therapy With Irbesartan and Atorvastatin.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IKPD 03-02
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-09-28 (Estimated); Status verified 2006-07

CONDITIONS: Healthy Subjects
Keywords: venoconstriction; venodilation; pleiotropic effects
MeSH Terms: interventions — Atorvastatin; Irbesartan

INTERVENTIONS:
Drug: atorvastatin
Drug: irbesartan

SUMMARY:
Vascular responses to angiotensin II and histamine are compared before and after 30 days of systemic treatment with either irbesartan 150 mg or atorvastatin 20 mg.

DETAILED DESCRIPTION:
Vascular responses to angiotensin II and histamine are compared before and after 30 days of systemic treatment with either irbesartan 150 mg or atorvastatin 20 mg.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* no relevant disease
* amendment: hypercholesterolaemic subjects

Exclusion Criteria:

* any relevant disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2003-03; Study Completion 2006-10

PRIMARY OUTCOMES:
vascular responses after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Kirch, MD, Study Chair — Institute of Clinical Pharmacology
Locations (1):
- Institute of Clinical Pharmacology, Medical Faculty, University of Technology, Dresden, Germany

REFERENCES:
- [Derived] Schindler C, Guenther K, Hermann C, Ferrario CM, Schroeder C, Haufe S, Jordan J, Kirch W. Statin treatment in hypercholesterolemic men does not attenuate angiotensin II-induced venoconstriction. PLoS One. 2014 Sep 29;9(9):e103909. doi: 10.1371/journal.pone.0103909. eCollection 2014. PMID 25264877